CLINICAL TRIAL: NCT00111111
Title: A Multicenter, Open-Label, Prospective Study to Evaluate the Effectiveness and Safety of Etanercept in the Treatment of Subjects With Psoriasis
Brief Title: An Evaluation of Etanercept in the Treatment of Subjects With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20030190
Record Dates: First submitted 2005-05-17; First posted 2005-05-18 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this multicenter, open-label, prospective study is to evaluate the effectiveness and safety of etanercept in the treatment of subjects with psoriasis.

ELIGIBILITY:
Inclusion Criteria: - Stable, active plaque psoriasis involving greater than or equal to 10% of body surface area (BSA) at screening and baseline Exclusion Criteria: - Any grade 3 or 4 adverse event or infection within 28 days before screening, or between the screening visit and study drug initiation - Evidence of skin conditions (e.g., eczema) other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis - Psoralen plus ultraviolet A radiation (PUVA), oral retinoids, cyclosporine, alefacept (Amevive®), efalizumab (Raptiva®), or any other systemic anti-psoriasis therapy within 28 days of study drug initiation - Ultraviolet light B (UVB) therapy, topical steroids, topical vitamin A or D analog preparations, or anthralin within 14 days of study drug initiation (exception: topical steroids, at no higher than moderate strength, are permitted on scalp, axillae, and groin but dose and formulation must remain stable throughout trial) - Prior exposure to any tumor necrosis factor (TNF)-inhibitor, including etanercept - Severe comorbidities - Known history of tuberculosis (TB), or previous positive purified protein derivative (PPD) test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Improvement in Physician's Global Assessment of Psoriasis

SECONDARY OUTCOMES:
Patient-reported outcomes including Dermatology Life Quality Index, SF-36, Euro-QoL 5D, and Beck Depression Index

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Moore A, Gordon KB, Kang S, Gottlieb A, Freundlich B, Xia HA, Stevens SR. A randomized, open-label trial of continuous versus interrupted etanercept therapy in the treatment of psoriasis. J Am Acad Dermatol. 2007 Apr;56(4):598-603. doi: 10.1016/j.jaad.2006.09.002. Epub 2006 Nov 17. PMID 17113190
- [Result] Gelfand JM, Kimball AB, Mostow EN, Chiou CF, Patel V, Xia HA, Freundlich B, Stevens SR. Patient-reported outcomes and health-care resource utilization in patients with psoriasis treated with etanercept: continuous versus interrupted treatment. Value Health. 2008 May-Jun;11(3):400-7. doi: 10.1111/j.1524-4733.2007.00251.x. PMID 18489665
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20030190.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com